CLINICAL TRIAL: NCT06377670
Title: Study of Functional and Aesthetic Outcomes After Wassel IV Thumb Duplication Surgery in Pediatric Population, With a Follow-up of at Least One Year
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC24.0012
Record Dates: First submitted 2024-03-05; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Wassel IV Thumb Duplication
Keywords: functional outcomes; aesthetic outcomes; pediatric surgery; thumb reconstruction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wassel IV Thumb Duplication Cases: This group consists of pediatric patients who have undergone surgical correction for Wassel IV thumb duplication. All participants have had a minimum of one year post-operative follow-up. This cohort will be assessed for functional and aesthetic outcomes using the Japanese Society for Surgery of the Hand (JSSH) scoring method. This includes evaluating thumb mobility, functionality, global aesthetics, and other quality of life aspects for each patient using their contralateral healthy thumb as a control. Data will be collected on preoperative metacarpophalangeal angle, type of skin flap used, surgical reconstruction technique, immobilization method, postoperative complications, and patient satisfaction with surgery and daily pain levels.
  Interventions: Procedure: Wassel IV Thumb Duplication Surgery

INTERVENTIONS:
Procedure: Wassel IV Thumb Duplication Surgery — This intervention involves the surgical correction of Wassel IV thumb duplication, which is a congenital hand anomaly. The study retrospectively evaluates the outcomes of various surgical techniques that have been employed to correct this condition, with a focus on functionality and aesthetics of the thumb post-surgery. Data collected post-intervention include preoperative metacarpophalangeal angle, type of skin flap, surgical reconstruction technique, immobilization method, and postoperative complications. Additionally, patient satisfaction and daily pain levels are assessed using standardized questionnaires. Each patient serves as their own control, with outcomes compared to their contralateral healthy thumb.

SUMMARY:
The purpose of this study is to evaluate the functional and aesthetic outcomes in children with Wassel IV thumb duplication

DETAILED DESCRIPTION:
Wassel IV thumb duplication is a congenital hand anomaly characterized by the presence of two adjacent thumbs. This condition has significant functional and aesthetic implications.

Previous studies have highlighted the complexity of the surgical management of Wassel IV thumb duplication, underscoring the need for an individualized approach for each case. Early interventions are often recommended to optimize long-term functional and aesthetic outcomes.

The field of study for evaluating these outcomes focuses on the analysis of the medium and long-term consequences of surgical interventions in children with this malformation. Evaluation criteria may include hand functionality, thumb mobility, overall aesthetics, and other aspects relevant to the quality of life of the affected pediatric patients. This medium and long-term approach offers crucial insights for refining treatment protocols and improving the overall management of this condition.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Wassel IV thumb duplication
* Pediatric patients aged between 1 and 18 years
* Minimum of one year post-operative follow-up
* Availability of radiographic, photographic, and medical data
* Regular post-operative medical follow-up with the referring surgeon
* Legal guardian and patient consent (non-opposition) to participate in the study

Exclusion Criteria:

* Subjects under guardianship or deprived of liberty
* Opposition from legal guardians or from the patient to participate in the study

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients who have undergone surgical correction for Wassel IV thumb duplication and have been followed up for at least one year post-surgery. The study population includes patients from the CHU Grenoble Alpes and Clinique Val d'Ouest Lyon.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-25 (Estimated); Primary Completion 2024-05-06 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Functional and Aesthetic Outcomes | Up to one year post-surgery for the primary outcome measure time frame
  Evaluation of functional and aesthetic outcomes using the Japanese Society for Surgery of the Hand (JSSH) scoring method. Functional outcomes include thumb mobility and function scored out of 10 points, and aesthetic outcomes include overall thumb appearance scored out of 14 points. The minimal and worst score is 0, the maximal and best score is 30.

SECONDARY OUTCOMES:
Comparison of Surgical Techniques | One year post-operative, to align with the follow-up period of the primary outcome measure.
  Evaluate which surgical reconstruction techniques yield better functional and aesthetic outcomes.
  Soft tissue reconstruction only or need for osteotomy.
Efficacy of Skin Flap Types | One year post-operative, to align with the follow-up period of the primary outcome measure.
  Assess the outcomes associated with different types of skin flaps used in the surgical correction.
  Number of "racquet skin plasty" and number of "Dautel flap". The evaluation of skin flaps will be assessed by various measures: the circumference of the thumb in millimeters, the appearance of the scar by self-assessment (visual analogue scale), and the symmetry of the thumb by self-assessment (visual analogue scale). All these measures are integrated into the JSSH score.
Immobilization Method Analysis | One year post-operative, to align with the follow-up period of the primary outcome measure.
  Determine the effectiveness of various immobilization methods post-surgery. Plaster immobilization or splint, with or without wire.
Preoperative Angle Decision Model | One year post-operative, to align with the follow-up period of the primary outcome measure.
  Measurement of the preoperative metacarpophalangeal angle of the thumb to be reconstructed.
  Develop a decision-making model for surgery based on the preoperative radiographic metacarpophalangeal angle.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dautel G, Perrin P. Use of an Axial Flap to Increase the Girth of Wassel IV Thumb Reconstructions. J Hand Surg Am. 2015 Jul;40(7):1327-32. doi: 10.1016/j.jhsa.2015.02.032. Epub 2015 Apr 16. PMID 25892712
- [Result] Luangjarmekorn P, Virojanawat N, Pongpacharaamphon P, Kitidumrongsook P. Preoperative angulation as a predictor for operations of Wassel type IV polydactyly. J Pediatr Orthop B. 2021 Nov 1;30(6):605-610. doi: 10.1097/BPB.0000000000000806. PMID 32956284
- [Result] Dijkman R, Selles R, van Rosmalen J, Hulsemann W, Mann M, Habenicht R, Hovius S, van Nieuwenhoven C. A clinically weighted approach to outcome assessment in radial polydactyly. J Hand Surg Eur Vol. 2016 Mar;41(3):265-74. doi: 10.1177/1753193415601336. Epub 2015 Aug 28. PMID 26319288
- [Result] Kayalar M, Gurbuz Y, Kucuk L, Sugun TS, Ademoglu Y, Ozaksar K. Surgical reconstruction in Wassel type IV thumb duplication. Acta Orthop Traumatol Turc. 2014;48(2):181-6. doi: 10.3944/AOTT.2014.13.0042. PMID 24747627